CLINICAL TRIAL: NCT00442858
Title: Incidence of Cardiovascular Diseases in Patients With Hypopituitarims
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Other Study IDs: LU-286-99
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Cardiovascular Diseases
Keywords: cardiac disease; cerebrovascular disease; GH deficiency; diabetes mellitus; hypertension; GH therapy; GH deficiency and hypopituitarims
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cerebrovascular Disorders; Dwarfism, Pituitary; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study was therefore two-fold: 1) to make a retrospective comparison of incidence of non-fatal stroke and cardiac events between a large cohort of patients with confirmed GHD on replacement therapy (including GH) and a control cohort from the general population; 2) to compare the prevalence of DM and cardioprotective medication between the cohorts at the time of questionnaire distribution with adjustment for possible confounders and effect modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed GH deficiency

Exclusion Criteria:

* Not confirmed GH deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800
Dates: Start 1999-01; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Eva Marie T Erfurth, MD, PhD, Principal Investigator — Endocrine Unit, Department of Medicine, University Hospital, Lund